CLINICAL TRIAL: NCT03541551
Title: Randomized Controlled Study to Evaluate Safety and Efficacy of Ologen® Collagen Matrix in Patients With Primary Congenital Glaucoma Undergoing Trabeculectomy
Brief Title: Ologen® Collagen Matrix in Patients With Primary Congenital Glaucoma Undergoing Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, HERF, Consultant-Ophthalmologist, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIS-90516
Record Dates: First submitted 2018-03-16; First posted 2018-05-30 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Primary Congenital Glaucoma; Developmental Glaucoma; Infantile Glaucoma
MeSH Terms: conditions — Hydrophthalmos | interventions — collagen-glycosaminoglycan copolymer; Trabeculectomy

STUDY DESIGN:
Intervention Model Description: Product:ologen® Collagen Matrix, Model: 830601, Shape:Round cylindrical, Size:6mm (diameter) x 2mm (thickness, Manufacturer: Aeon Astron Europe B. V.
Who Masked: Participant, Investigator
Masking Description: Eligible patient after screening will be assigned consecutive randomization numbers in ascending order upon enrollment. The patient will be randomized in 1:1ratio to one of two study groups, namely combined trabeculotomy with trabeculectomy with ologen® Collagen Matrix as adjunctive wound modulator(Group A) or combined trabeculotomy with trabeculectomy alone without any adjunctive (Group B). The assigned randomization number will be recorded in each subject's DCF. The randomization scheme will be generated using random function in excel before patient enrollment in order to avoid investigator's patient selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTT with ologen® Collagen Matrix (Experimental): Experimental: Trabeculotomy with trabeculectomy with ologen implant
  Interventions: Procedure: CTT with ologen® Collagen Matrix
- Trab Trab (Active Comparator): Active Comparator: Trabeculotomy with trabeculectomy
  Interventions: Procedure: Trab Trab

INTERVENTIONS:
Procedure: CTT with ologen® Collagen Matrix — ologen® Collagen Matrix approved by Indian health authority with registration numberof MD-1517 will be provided by Aeon Ajanta India Pvt. Ltd. free of cost for this clinical research only.
  Other Names: Ologen with combined trabeculotomy and trabeculectomy
  Arms: CTT with ologen® Collagen Matrix
Procedure: Trab Trab — combined trabeculotomy with trabeculectomy
  Other Names: combined trabeculotomy with trabeculectomy
  Arms: Trab Trab

SUMMARY:
To the best of Investigator knowledge, no studies to this date have compared the safety and efficacy of ologen® Collagen Matrix in Primary congenital glaucoma (PCG) patients undergoing trabeculectomy. Given that filtration surgery is usually less successful in patients with developmental glaucoma; the purpose of this study is to compare combined trabeculectomy with trabeculotomy (CTT) with adjuvant ologen® Collagen Matrix versus CTT without ologen® in children with PCG. Investigator hypothesis is that CTT with ologen® Collagen Matrix would be as effective as CTT in IOP control, but with reduced scarring and long term healthier bleb morphology.

DETAILED DESCRIPTION:
Standard combined trabeculectomy with trabeculotomy (CTT) All CTT surgeries will be performed under general anesthesia.Under aseptic surgical technique, a superior rectus suture will be placed using 4'0 silk and a limbal-based conjunctival flap to be performed. Sub-Tenon dissection and hemostasis will be achieved and a half-thickness 4 x 4mm rectangular scleralflap will to be dissected up to clear cornea, and radial incision will be placed at the location of the schemes canal, Harms trabepculotome will be used to pass into the schemes canal and rotated into the anterior chamber to open app 60 degree on either sides, A 2 × 2 mm deep scleral block will be excised and peripheral iridectomy will be performed. The scleral flap will be closed with one 10-0 nylon suture and conjunctiva will be closed with 8-0 vicryl continuous suture.

The same procedure will be done for the CTT with ologen® except, before closing the conjunctiva, the ologen® implant will be placed subconjunctivally just overlapping the apex of the triangular scleral flap

ologen® Collagen Matrix ologen® Collagen Matrix approved by Indian health authority with registration numberof MD-1517 (valid till Mar-15-2018) will be provided by Aeon Ajanta India Pvt. Ltd. free of cost for this clinical research only.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month to 3 years (inclusive)
* Any case diagnosed as congenital glaucoma (with enlarged corneal diameter more than 11 mm, including corneal edema or Haab'sstria with or without optic disc cupping, IOP>12 mm Hg)
* Parents of the patientis willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

* Patients withany other types of secondary glaucoma
* Patients with any other ocular disease

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Comparing IOP control between the two groups:Change of intraocular pressure (IOP) over time | 12 months
  Assess control of IOP over time. "Complete success" is defined as IOP reduction of >20% and / or an IOP constantly <21 mmHg without any antiglaucoma medication. "Qualified success" is defined as IOP < 21 mmHg with topical antiglaucoma medication. "Failure" is defined as IOP > 21mmHg in 2 subsequent follow visits despite topical antiglaucoma medication.

SECONDARY OUTCOMES:
Comparing bleb morphology in two groups by change of Moorfields Bleb Grading System (MBGS) score over time | 12 months
  Assess bleb characteristics using Moorfields Bleb Grading System (MBGS) score as measurement tool to document bleb grading score over time, clinically and with photographs

CONTACTS AND LOCATIONS:
Overall Officials: senthil sirisha, MS, Principal Investigator — YES
Locations (1):
- Charitha, Hyderabad, Telangana, India